CLINICAL TRIAL: NCT04262661
Title: A Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneous NNC0472-0147 in Healthy Subjects and in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Look at How Safe NNC0472-0147 is in Healthy People and in People With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1147-4527; U1111-1232-3957 (Other: World Health Organization (WHO)); 2019-001927-11 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Healthy Volunteers; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Intervention Model Description: Part 1: Single ascending dose, placebo control. Part 2: Multiple ascending dose design, active control.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NNC0472-0147 Part 1 (Experimental): Part 1: Each cohort will consist of 8 healthy subjects - 6 subjects will receive a single subcutaneous (s.c., under the skin) dose of NNC0472-0147.
  Interventions: Drug: NNC0472-0147
- Placebo Part 1 (Placebo Comparator): Part 1: Each cohort will consist of 8 healthy subjects - 2 subjects will receive a single s.c. dose of placebo.
  Interventions: Drug: Placebo (NNC0472-0147)
- NNC0472-0147 Part 2 (Experimental): Part 2: Each cohort will consist of 12 subjects with T2DM. 9 subjects will receive once daily s.c. doses of NNC0472-0147 for 14 days
  Interventions: Drug: NNC0472-0147
- Insulin glargine Part 2 (Active Comparator): Part 2: Each cohort will consist of 12 subjects with T2DM - 3 subjects will receive once daily s.c. doses of insulin glargine for 14 days.
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: NNC0472-0147 — Part 1: A single dose of NNC0472-0147, dose increased in each cohort. Part 2: Daily doses of NNC0472-0147, dose increased in each cohort.
  Arms: NNC0472-0147 Part 1; NNC0472-0147 Part 2
Drug: insulin glargine — Part 2: A fixed dose level of 0.5 U/kg insulin glargine will be used in all cohorts.
  Arms: Insulin glargine Part 2
Drug: Placebo (NNC0472-0147) — Part 1: A single dose of placebo, dose increased in each cohort.
  Arms: Placebo Part 1

SUMMARY:
This study is investigating the safety and tolerability of the new medicine NNC0472-0147, its concentrations in the blood and its effect on blood sugar for the treatment of diabetes. Another goal of the study is to determine an effect of NNC0472-0147 on cholesterol. The first part of the study is conducted in healthy people, while the second part involves people with type 2 diabetes (T2DM). The study will test how NNC0472-0147 is tolerated by the body, how it is taken up in the blood, how long it stays there and how much blood sugar is lowered. In part 1, participants will either get the new medicine NNC0472-0147 or placebo (an injection that does not contain active medicine) - which treatment is decided by chance. In part 2, participants will either get the new medicine NNC0472-0147 or insulin glargine - which treatment is decided by chance. It is the first time that NNC0472-0147 is tested in humans. Participants will get once daily injections of either NNC0472-0147 or insulin glargine for a treatment period of fourteen days. The injections will be given under the skin (subcutaneously, s.c.) of the left thigh. Participants will be in the study for about 7 weeks. There will be 15 visits with the study doctor. People cannot be in the study if the study doctor thinks that there are risks for their health. Only women who cannot become pregnant are allowed to participate.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Male
* Aged 18-55 years (both inclusive) at the time of signing nformed consent.

Part 2:

* Male, or female of non-child bearing potential. Non-child bearing potential is defined by being surgically sterilised (documented hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or being postmenopausal (no menses for 12 months without an alternative medical cause) prior to the day of screening.
* Aged 18-64 years (both inclusive) at the time of signing informed consent.
* Diagnosed with T2DM at least 180 days prior to the day of screening.
* Treated with any insulin for 90 days or longer prior to the day of screening.
* Low-density lipoprotein cholesterol level above 1.80 mmol L.

Exclusion Criteria:

Part 1:

- Male of reproductive age who or whose partner(s) is not using highly effective contraceptive methods (highly effective contraceptive measures as required by local regulation or practice). Highly effective contraceptive measures include that the male subject uses a condom during intercourse and that the partner practices highly effective contraception (risk of pregnancy must be lower than 1%). In addition, subjects must not donate sperm for the duration of the trial.

Part 2:

* Male of reproductive age who or whose partner(s) is not using highly effective contraceptive methods (highly effective contraceptive measures as required by local regulation or practice). Highly effective contraceptive measures include that the male subject uses a condom during intercourse and that the partner practices highly effective contraception (risk of pregnancy must be lower than 1%). In addition, subjects must not donate sperm for the duration of the trial.
* Use of oral antidiabetic drugs (OADs) other than metformin or use of glucagon-like peptide-1 (GLP-1) receptor agonists (e.g. exenatide, liraglutide, semaglutide) within 90 days prior to the day of screening.
* Treatment with peptide proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors within 180 days prior to the day of screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of treatment emergent adverse events | From IMP administration at day 1 (visit 2) until completion of post-treatment end-of-trial visit (day 15, visit 6)
  Number of events
Part 2: Number of treatment emergent adverse events | From IMP administration at day 1 (visit 2) until completion of post-treatment end-of-trial visit (day 30, visit 14)
  Number of events

SECONDARY OUTCOMES:
Number of hypoglycaemic episodes of alert value (level 1) below 3.9 mmol/L (70 mg/dL) and equal to or above 3.0 mmol/L (54 mg/dL) | From IMP administration at day 1 (visit 2) until completion of post-treatment end-of-trial visit (day 15, visit 6)
  Number of episodes
Number of hypoglycaemic episodes of alert value (level 1) below 3.9 mmol/L (70 mg/dL) and equal to or above 3.0 mmol/L (54 mg/dL) | From IMP administration at day 1 (visit 2) until completion of post-treatment end-of-trial visit (day 30, visit 14)
  Number of episodes
Number of clinically significant hypoglycaemic episodes (level 2) below 3.0 mmol/L (54 mg/dL) | From IMP administration at day 1 (visit 2) until completion of post-treatment end-of-trial visit (day 15, visit 6)
  Number of episodes
Number of clinically significant hypoglycaemic episodes (level 2) below 3.0 mmol/L (54 mg/dL) | From IMP administration at day 1 (visit 2) until completion of post-treatment end-of-trial visit (day 30, visit 14)
  Number of episodes
Number of severe hypoglycaemic episodes (level 3) | From IMP administration at day 1 (visit 2) until completion of post-treatment end-of-trial visit (day 15, visit 6)
  Number of episodes
Number of severe hypoglycaemic episodes (level 3) | From IMP administration at day 1 (visit 2) until completion of post-treatment end-of-trial visit (day 30, visit 14)
  Number of episodes
Area under the serum NNC0472-0147 concentration-time curve after a single dose | From 0 hours until infinity after a single IMP administration at day 1 (visit 2).
  pmol*h/L
Maximum observed serum NNC0472-0147 concentration after a single dose | From 0 hours until last measurement time after a single IMP administration at day 1 (visit 2)
  pmol/L
Area under the serum NNC0472-0147 concentration-time curve during one dosing interval at steady state | From 0 to 24 hours after last multiple IMP administration at day 14 (visit 9)
  pmol*h/L
Maximum observed serum NNC0472-0147 concentration at steady state | From 0 to 24 hours after last multiple IMP administration at day 14 (visit 9)
  pmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor & Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (2):
- Germany (2):
  - Novo Nordisk Investigational Site, Mainz
  - Novo Nordisk Investigational Site, Neuss

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com